CLINICAL TRIAL: NCT00488423
Title: Glucose Metabolism in the Immediate and Short Term Follow up From Bariatric Surgery
Brief Title: Glucose Metabolism in the Immediate and Short Term Follow up After Bariatric Surgery
Acronym: MIDAS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Ethicon Endo-Surgery (Industry)
Responsible Party: Cleveland Clinic Foundation, Endocrine & Metabolic Institute Research
Allocation: Non-Randomized | Model: Single Group | Masking: Single
Other Study IDs: 8585; NCT00554593 (obsolete NCT alias)
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes; Gastric Bypass
Keywords: diabetes; MIDAS; gut hormones; gastric bypass; lap band
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lap-band (Active Comparator): Patient undergoing Lap-band Bariatric Surgery
  Interventions: Procedure: Mixed Meal Tolerance test, Hyperglycemic clamp
- Gastric Bypass (Active Comparator): Patient's undergoing Laparoscopic Roux-N Y Gastric Bypass surgery.
  Interventions: Procedure: Mixed Meal Tolerance test, Hyperglycemic clamp

INTERVENTIONS:
Procedure: Mixed Meal Tolerance test, Hyperglycemic clamp — Subjects undergo a standard mixed meal tolerance test & hyperglycemic clamp to assess insulin secretion & sensitivity (whole body glucose disposal) pre-op. Following surgery, at 1week, 1 month, 6 months and 12 months subjects will undergo hyperglycemic clamp & mixed meal tolerance test. During these tests, measurements will include plasma levels of glucose, insulin, C-peptide, free fatty acid levels and adipocyte hormone profile (adiponectin, leptin, resistin). A gut hormone profile (ghrelin, glucagons-like-peptide 1 GLP-1, glucose-dependent insulinotropic polypeptide GIP, PYY) will be performed at fasting & specific postprandial times. Results will be compared between two groups: patients undergoing laparoscopic Roux-en-Y gastric bypass & gastric banding.
  Other Names: MMTT

SUMMARY:
MIDAS involves an assessment of glucose levels obtained before and after bariatric surgery. There are two different procedural tests involved; an oral glucose tolerance test (mixed meal) and a hyperglycemic clamp test. Two tests are performed preoperatively and five more are performed postoperatively for a one year period. The associated labwork drawn with the mixed meal and clamp tests are demonstrating changes in glucose, insulin and gut hormone levels.

DETAILED DESCRIPTION:
Tests performed are the Mixed Meal tolerance test, the Hyperglycemic Clamp test, c-peptide, free fatty acids, adipocyte hormone profile levels.

ELIGIBILITY:
Inclusion Criteria:

* Negative pregnancy test if female
* ADA criteria for diabetes type II
* Hematocrit > 35 creatinine < 1.9, AST < 3X upper limit of normal, ALT < 3X upper limit of normal, alkaline phos <3X upper limit of normal
* Eligibility for bariatric surgery based on the NIH and clinical criteria
* Mentally and legally capable of providing consent

Exclusion Criteria:

* Lactating females
* Must not have type I diabetes
* Systemic steroids taken within 6 months
* Clinically significant heart disease
* Recent pulmonary embolism, untreated proliferative retinopathy, renal failure, uncontrolled hypertension, autonomic neuropathy, resting heart rate > 100, neuromuscular or musculoskeletal disease.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2006-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To assess the effect of gastric by-pass surgery to decrease lipotoxicity. | One year

SECONDARY OUTCOMES:
To examine the effect of roux-en-Y compared to gastric banding on pancreatic B cell recovery or insulin secretion in response to oral and IV glucose. | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Sangeeta R. Kashyap, MD, Principal Investigator — The Cleveland Clinic; Philip R. Schauer, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States